CLINICAL TRIAL: NCT01355549
Title: A Pilot Study to Evaluate the Feasibility of Platelet-Rich Plasma Therapy as a Treatment for Chronic Shoulder Pain in Persons With Spinal Cord Injury
Brief Title: Platelet-Rich Plasma Therapy for Shoulder Pain in Persons With Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Trevor Dyson-Hudson, M.D., Interim-Director, Spinal Cord Injury Research, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-677-10
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Shoulder Pain; Rotator Cuff Tendinitis; Rotator Cuff Syndrome; Spinal Cord Injury
Keywords: Shoulder pain; Rotator cuff disease; Spinal cord injuries; Platelet-rich plasma therapy; Rehabilitation
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries; Spinal Cord Injuries | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet-rich plasma therapy (Experimental): Platelet rich plasma (PRP) describes a new technology in which platelets are isolated from a sample of a person's own blood using simple cell-separating systems such as centrifugation in order to obtain highly concentrated samples of platelets that can be re-injected into an injury site to promote healing.
  Interventions: Biological: Platelet-rich plasma (PRP) therapy

INTERVENTIONS:
Biological: Platelet-rich plasma (PRP) therapy — Platelet rich plasma (PRP) describes a new technology in which platelets are isolated from a sample of a person's own blood using simple cell-separating systems such as centrifugation in order to obtain highly concentrated samples of platelets that can be re-injected into an injury site to promote healing.
  Other Names: Autologous blood injections

SUMMARY:
Shoulder pain is common in persons with spinal cord injury (SCI). It is most often caused by overuse injuries to the muscles and tendons that can occur during wheelchair propulsion, transfers, and other activities of daily living. Normally, shoulder pain resolves with conservative treatments such non-steroidal anti-inflammatory drugs (e.g. aspirin, ibuprofen, naproxen, etc.) and physical therapy. However, when these treatments fail, shoulder surgery may be the only option.

Platelet Rich Plasma therapy, or PRP, is a treatment option for non-healing muscle and tendon injuries such as those that cause shoulder pain in persons with SCI. Using one's own blood, cells within the blood called "platelets" are concentrated and then re-injected into the muscle and tendon of the shoulder. These platelets release substances known as "growth factors" that lead to tissue healing. By concentrating the platelets we increase the growth factors up to eight times which will promote the healing of tendons. PRP therapy has shown promise in treating tendon and muscle injuries in able-bodied persons; however, its effectiveness in persons with SCI is unknown. The purpose of this study is to explore the feasibility, safety, and efficacy of PRP therapy for chronic shoulder pain in persons with SCI. The human body has a remarkable ability to heal itself and we hypothesize that re-injecting concentrated platelets will facilitate the natural healing process and will reduce shoulder pain in persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, 18 to 60 years of age, inclusive.
* The subject has neurological impairment secondary to a spinal cord injury that occurred at least twelve (12) months prior to the Screening Visit and the level of the injury is between C6 and L5, inclusive.
* The subject is non-ambulatory except for exercise purposes and uses a manual or power wheelchair as his/her primary means of mobility (> 40 hours/week).
* The subject currently has chronic shoulder pain due to rotator cuff disease in spite of at least 6 months of conservative treatment. Average shoulder pain intensity during the week leading up to the Screening Visit should be at least 5 out of 10 on an 11-point numerical rating scale (NRS; 0, no pain; 10, maximum pain imaginable), in spite of a past history of completing 6 months of conservative treatment. Rotator cuff disease will be defined as pain over the anterior shoulder, with direct palpation and pain at the shoulder with provocative tests for rotator cuff disease that is confirmed by tendinopathic changes on ultrasound imaging.
* The subject is able and willing to comply with the protocol.
* The subject is able to and has voluntarily given informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* The subject reports prior PRP treatment in the same shoulder;
* The subject reports a history of systemic disorders, such as diabetes or rheumatoid arthritis;
* The subject has contra-indications to the procedure, such as infection, coagulopathy, or is currently taking anti-coagulants;
* The subject reports having a glucocorticoid injection in the past 4 weeks;
* The subject is pregnant (documented by a urine pregnancy test);
* The subject has any medical condition, including psychiatric disease, which would interfere with the interpretation of the study results or the conduct of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the PRP treatment.
  Shoulder pain intensity will also be assessed weekly using a numerical rating scale (NRS). Subjects will be asked to rate their average pain, most severe pain, and least severe pain during the past week using an 11-point scale (i.e. 0-10) anchored at the ends by "no pain" and "worst pain ever experienced." An 11-point NRS measure of pain intensity allows for comparison across clinical trials of chronic pain treatment and is recommended as a core outcome measure for chronic pain clinical trials.

SECONDARY OUTCOMES:
Wheelchair User's Shoulder Pain Index (WUSPI) | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the PRP treatment.
  The WUSPI is a 15-item self-report instrument that measures shoulder pain intensity in wheelchair users during various ADLs, such as transfers, loading a wheelchair into a car, wheelchair mobility, dressing, bathing, overhead lifting, driving, performing household chores, and sleeping. Each item is scored using a 10cm visual analog scale (VAS) which is anchored at the ends with "no pain" and "worst pain ever experienced." Individual item scores are summed to arrive at a total index score, which ranges from 0 to 150.
Patient Global Impression of Change | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the PRP treatment.
  Subjects will be asked to rate on a 7-point scale overall impression following treatment as compared to the previous measurement interval. The 7-point PGIC scale (anchored by "very much improved" and "very much worse") is used to measure global treatment effect.
Brief Pain Inventory interference items (BPI-I) | Baseline and 4 weeks, 8 weeks, 12 weeks, and 24 weeks after the PRP treatment.
  The Brief Pain Inventory (BPI) was developed by Cleeland, and has been used in a number of investigations of chronic pain. Its pain interference subscale has been used in several investigations of pain in SCI. In its original version the subscale (BPI-I7) consisted of 7 items measuring interference with general activity, sleep, mood, relationships, etc.). For uses with an SCI sample, in item 3 of BPI-I7, ''walking ability'' is replaced by "ability to get around."
Rotator Cuff Disease Score | Baseline and at the 12-Week and 24-Weeks Follow-up Visit after the PRP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor A. Dyson-Hudson, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

REFERENCES:
- [Derived] Dyson-Hudson TA, Hogaboom NS, Nakamura R, Terry A, Malanga GA. Ultrasound-guided platelet-rich plasma injection for the treatment of recalcitrant rotator cuff disease in wheelchair users with spinal cord injury: A pilot study. J Spinal Cord Med. 2022 Jan;45(1):42-48. doi: 10.1080/10790268.2020.1754676. Epub 2020 May 7. PMID 32379581